CLINICAL TRIAL: NCT01324778
Title: An Open, Randomized, Prospective Multi Centre Study Comparing OsseoSpeedTM TX With OsseoSpeedTM in the Partially and Totally Edentulous Maxillae
Brief Title: Multi Centre Study Comparing OsseoSpeed TX With OsseoSpeed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YA-OTX-0001
Record Dates: First submitted 2011-03-22; First posted 2011-03-29 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Partial Edentulism; Edentulism Nos
Keywords: Edentulism in the Upper Jaw

ARMS (2):
- A (Experimental)
  Interventions: Device: OsseoSpeed TX
- B (Active Comparator)
  Interventions: Device: OsseoSpeed

INTERVENTIONS:
Device: OsseoSpeed TX — OsseoSpeedTM TX implants of lengths 6-17 mm
  Arms: A
Device: OsseoSpeed — OsseoSpeedTM implants of lengths 6-17 mm
  Arms: B

SUMMARY:
To compare marginal bone level alterations, implant stability and implant survival between OsseoSpeed och OsseoSpeed TX

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent
2. Female/male aged 18 years and over
3. History of edentulism in the study area of at least 3 months
4. In need for implant(s) replacing missing tooth/teeth in the maxilla
5. Deemed by the investigator to be suitable for one stage surgery
6. Deemed by the investigator to be suitable for loading after 10-12 weeks
7. Deemed by the investigator as likely to present an initially stable implant situation.
8. Deemed by the investigator to have a "functional" opposing dentition at the time of loading the implants.

Exclusion criteria:

1. Unlikely to be able to comply with study procedures, as judged by the investigator
2. Uncontrolled pathological processes in the oral cavity
3. Known or suspected current malignancy
4. History of radiation therapy in the head and neck region
5. History of chemotherapy within 5 years prior to surgery
6. Systemic or local disease or condition that would compromise post-operative healing and/or osseointegration
7. Uncontrolled diabetes mellitus
8. Corticosteroids or any other medication that would compromise post-operative healing and/or osseointegration
9. Present alcohol and/or drug abuse
10. Current need for bone grafting and/or augmentation in the planned implant area
11. Involvement in the planning and conduct of the study (applies to both Astra Tech staff and staff at the study site)
12. Previous enrolment in the present study.
13. Simultaneous participation in another clinical study, or participation in a clinical study during the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2011-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Marginal Bone Level | One year after loading
  Marginal Bone Level will be determined from radiographs and expressed as the difference from a reference point on the implant to the most coronal bone-to-implant contact on the mesial and distal aspect of the implant. Marginal Bone Level expressed in millimeters at the 12 months follow-up visit will be compared to values obtained at delivery of permanent restoration i.e. loading (baseline).

SECONDARY OUTCOMES:
Implant stability | At implant placement (inclusion) (day 1)
  Implant stability will be evaluated clinically/manually (recorded as stable yes/no)
Implant stability | At implant placement (inclusion) (day 1)
  Implant stability will be evaluated using Resonance Frequency Analysis (RFA)
Implant stability | At implant loading (10-12 weeks after implant placement)
  Implant stability will be evaluated clinically/manually (recorded as stable yes/no)
Implant survival | One year after loading
  Implant survival rate will be evaluated by clinically and radiographically counting the number of remaining implants from implant placement to one year after loading.

CONTACTS AND LOCATIONS:
Overall Officials: Carl-Johan Ivanoff, DDS, PhD, Principal Investigator — Colosseumkliniken Mölndal
Locations (11):
- Sweden (11):
  - Specialisttandvården, Hallands sjukhus, Halmstad
  - Avd. för Parodontologi / Avd. för Oral Protetik, Odontologiska Institutionen, Jönköping
  - Specialist- och sjukhustandvården, Kalmar
  - Centrum för Oral Rehablilitering, Linköping
  - Colossseumkliniken Mölndal, Mölndal
  - Käkkirurgiska kliniken / Protetikkliniken, Örebro
  - Käkcentrum, Södersjukhuset, Stockholm
  - Specialisttandvården, S:t Eriks Sjukhus, Stockholm
  - Käkkirurgiska kliniken NÄL / Specialistcentrum Uddevalla sjukhus, Trollhättan
  - Käkkirurgiska Kliniken/Protetikkliniken, Umeå
  - Parodontologi kliniken och Protetik- och Bettfysiologiska kliniken, Vaxjo

REFERENCES:
- [Derived] Ivanoff CJ, Lindhe J, Ellner S, Johansson KJ, Abrahamsson P. An open, randomised, multi-centre study, comparing straight and tapered apex implants design, in partially and totally edentulous maxillae. Acta Odontol Scand. 2021 Oct;79(7):492-498. doi: 10.1080/00016357.2021.1894352. Epub 2021 Mar 5. PMID 33666125